CLINICAL TRIAL: NCT07093723
Title: Protein S100B Versus Neutrophils/Lymphocytes Ratio in Early Prediction of Brain Injury
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Asmaa Mahmoud Abdel Hamid Elmesiry, Lecturer of Pediatrics, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Other Study IDs: 36264PR392/10/23
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: S100B; Neutrophils/Lymphocytes Ratio; Prediction; Brain Injury
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Preterm neonates, their gestational age between 28- 36 gestational weeks
  Interventions: Diagnostic Test: S100B Protein; Diagnostic Test: Neutrophils to Lymphocytes ratio

INTERVENTIONS:
Diagnostic Test: S100B Protein — Serum level of S100B Protein was measured on the first and third days of seizure activity by ELISA.
Diagnostic Test: Neutrophils to Lymphocytes ratio — Neutrophils to Lymphocytes ratio was measured on the first and third day of seizure activity obtained by complete blood count.

SUMMARY:
The study aimed to evaluate the role of Protein S100B versus the neutrophil-to-lymphocyte ratio (NLR) as an early predictor biomarker and the value of amplitude-integrated electroencephalography (aEEG) as an early predictor and prognostic method for neonatal brain injury susceptibility and severity.

DETAILED DESCRIPTION:
The most prevalent types of newborn brain injury (NBI) are intraventricular haemorrhage (IVH), periventricular leukomalacia (PVL), and hypoxic-ischemic encephalopathy (HIE), which can affect neonates born at any gestational age (GA).

Amplitude-integrated EEG (aEEG) is another early predictor and prognostic technique for Neonatal Brain Injury. Electrophysiological brain activity, as measured by aEEG, is a well-established method for giving information on the functional and metabolic status of the brain and the incidence of epileptic seizure episodes.

S100B belongs to the S100 family. Because it is soluble in a 100% saturated solution of ammonium sulfate, it was designated "S100." S100 protein is a calcium-binding cytosolic protein with a molecular weight of 21 kDa comprised of 2 monomers, which are found in a variety of cells and are primarily concentrated in the glial cells of the CNS. Due to its molecular weight, peripheral blood will detect only S100B.

The neutrophil-to-lymphocyte ratio (NLR) reflects changes in neutrophil and lymphocyte levels, which is an indication of inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 28 and 36 weeks.
* Prematurity.

Exclusion Criteria:

* Intrauterine growth restriction (IUGR).
* Multiple congenital anomalies.
* Chromosomal abnormalities.
* Preterm less than 28 weeks.
* Infant of diabetic mother.

Ages: 28 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This prospective cross-sectional study will be conducted at the Neonatal Intensive Care Unit (NICU) of the Pediatric Department at Tanta University Hospitals over 3 months, from September 2023 to March 2024.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Protein S100B | Third day of seizure activity
  Serum level of S100B Protein was measured on the first and third days of seizure activity by ELISA.

SECONDARY OUTCOMES:
Neutrophils/Lymphocytes Ratio | Third day of seizure activity
  Neutrophils to Lymphocytes ratio was measured on the first and third day of seizure activity obtained by complete blood count.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.